CLINICAL TRIAL: NCT00710853
Title: Effects of Qigong, Tai Chi and Yog Practice on Indicators of Health and Quality of Life in Older Adults
Brief Title: Effects of Qigong, Tai Chi and Yoga Practice in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bastyr University (Other)
Collaborators: Gencare Incorporated (Industry)
Responsible Party: Wendy Weber, ND, MPH, PhD until 3/20/9 Mark Martzen, PhD thereafter, Bastyr University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: GC23B11
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: Geriatric; Qi gong; Yoga; Tai chi; Geriatric Assessment
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): YiRen Qi gong weekly class for 8 weeks
  Interventions: Other: YiRen Qi gong
- 2 (Experimental): Tai Chi weekly class for 8 weeks
  Interventions: Other: Tai Chi
- 3 (Active Comparator): Hatha yoga weekly class for 8 weeks
  Interventions: Other: Hatha yoga

INTERVENTIONS:
Other: YiRen Qi gong — One hour weekly class for 8 week duration
  Arms: 1
Other: Tai Chi — One hour weekly class for 8 week duration
  Arms: 2
Other: Hatha yoga — One hour weekly class for 8 week duration
  Arms: 3

SUMMARY:
The purpose of this study is to compare the effects of an 8-week intervention using YiRen Qigong, Tai Chi or Hatha yoga in older adults (age 70 and above) residing at a Gencare senior living facility. Outcome measures completed at the beginning and end of each intervention period will be blood pressure, heart rate, perceived quality of life (PQOL)and a symptoms questionnaire (SF-36), ability and speed of walking 20 feet (for ambulatory participants), and neck and arm range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Be a resident of a Gencare Senior Living facility in Granite Falls, Lynnwood, Renton, Ballard and Lake City, WA
* Be at least 70 years of age
* Be willing to participate in the tai chi, qi gong and/or yoga classes
* Willing to complete study-related outcomes assessments

Exclusion Criteria:

* Not medically able to participate in the mild level of activity involved in the 3 interventions as determined by the resident's physician
* Unable to complete study questionnaires or study procedures at screening

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure | End of 8-week class
Heart rate | End of 8-week class
Quality of life (SF-36 and PQOL) | End of 8-week class

SECONDARY OUTCOMES:
Adverse events | End of 8-week class

CONTACTS AND LOCATIONS:
Overall Officials: Mark Martzen, PhD, Principal Investigator — Bastyr University
Locations (3):
- United States (3):
  - Gencare-The Village at Granite Falls, Granite Falls, Washington
  - Gencare-Scriber Gardens, Lynnwood, Washington
  - Gencare-The Lodge at Eagle Ridge, Renton, Washington